CLINICAL TRIAL: NCT03966274
Title: A Prospective Multicenter Clinical Validation Study of DeltaScan for the Assessment of Delirium in the Intensive Care Unit and on Wards
Brief Title: DeltaScan Validation Study for the Assessment of Delirium in the ICU and on Wards
Acronym: Val3
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Radboud University Medical Center (Other); Tergooi Hospital (Other); Franciscus Gasthuis (Other); Erasmus Medical Center (Other); Isala (Other); OLVG (Network); St. Antonius Hospital (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Diakonessenhuis, Utrecht (Other); Amphia Hospital (Other); Prolira (Industry); European Union (Other)
Responsible Party: Principal Investigator, A.J.C. Slooter, Professor of Intensive Care Neuropsychiatry, UMC Utrecht
Other Study IDs: 17-857/C
Record Dates: First submitted 2019-04-05; First posted 2019-05-29 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Delirium
Keywords: Electroencephalography; Acute Confusion; Neurobehavioral Manifestations; Encephalopathy; Neurocognitive Disorders; Mental Disorders; Acute Brain Failure
MeSH Terms: conditions — Delirium; Neurobehavioral Manifestations; Brain Diseases; Neurocognitive Disorders; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirium positive
- Delirium negative

SUMMARY:
Rationale: Delirium is associated with prolonged hospitalization, an increased risk of dementia, institutionalization and mortality, as well as increased costs. Early detection of delirium would allow for early treatment and improved patient outcomes, but delirium is often not recognized and treatment is therefore delayed or not applied at all. Additionally, current screening tools are subjective, so an alternative, more objective diagnostic tool for early delirium detection is desired.

Objective: To investigate the diagnostic performance of the DeltaScan, a CE-certified device to detect delirium using a brief electroencephalography (EEG) recording. A single EEG recording will be obtained from patients admitted to an Intensive Care Unit (ICU), and elderly patient admitted to the ward.

Study design: Cross-sectional, multicenter study.

Study population: Adult patients admitted to an ICU, and elderly at the ward.

Main study parameters/endpoints: (1) Delirium as assessed by an adjudication committee of three delirium experts, based on cognitive information that is collected by one experienced investigator in line with the Diagnostic and Statistical Manual of Mental Disorders, 5th edition, (DSM-5) criteria (2) Delirium Probability as determined by DeltaScan, (3) the proportion of successful DeltaScan measurements, and (4) the repeatability of the DeltaScan measurements.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The burden to participants of this study is minimal. EEG recording using the CE-certified DeltaScan will be made using a strip with EEG electrodes that will be mounted to the head using self-adhesive gel. The patient will be visited by an experienced investigator, who collects information in accordance with DSM-5 criteria for delirium. This assessment will be performed once and takes about 10 minutes. Afterwards, the EEG recording will be performed once and takes a maximum of 4 minutes, and all procedures combined will take a maximum of 6-7 minutes. Both the EEG recording and the assessment are an add-on to routine care and will be performed within 30 minutes of each other.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the ICU or ward ICU patients: Richmond Agitation-Sedation Scale (RASS) score of -2 or higher Ward patients: aged 70 years or older
* Per the Instructions of Use of DeltaScan the patient has to be continuously awake at the time of the EEG measurement

Exclusion Criteria:

* Age younger than 18 years.
* Acute macro brain injury in 6 weeks prior to the DeltaScan measurement (such as postanoxic encephalopathy or traumatic brain injury).
* Admitted because of a primary neurological or neurosurgical disease
* Patients with severe agitation hampering measurement with DeltaScan.
* Patients who cannot clinically be assessed for delirium, e.g. due to a language barrier or deafness.
* Patients using lithium
* Patients with a metal plate or a metal device in the head
* Known pre-existing dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU or the ward
Sampling Method: Non-Probability Sample
Enrollment: 434 (Actual)
Dates: Start 2019-02-16 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
The positive and negative predictive value of DeltaScan | The predictive value of DeltaScan is assessed through study completion. Each patient is assessed only once, at a random time between admission and discharge to the ICU/nursing ward, for a maximum of 1 day.
  Using positive and negative predictive values, the diagnostic performance of the DeltaScan will be assessed separately in patients admitted to an ICU, and elderly patients admitted to the ward.
  A specific focus will be on a high negative predictive value (NPV) because it is important not to miss delirium. A lower positive predictive value (PPV) is acceptable, as the subsequent step in the management of patients with a positive Delta scan will be further diagnostic testing, which is clinically considered to have a lower risk compared to missed delirium.

SECONDARY OUTCOMES:
Sensitivity and Specificity of DeltaScan | Sensitivity and Specificity of DeltaScan is assessed through study completion. Each patient is assessed only once, at a random time between admission and discharge to the ICU/nursing ward, for a maximum of 1 day.
  To investigate the diagnostic performance in terms of sensitivity and specificity of the DeltaScan, separately in patients admitted to an ICU, and elderly patients admitted to a ward.
Proportion of successful DeltaScan measurements | From date of study start until the date of study completion. Each patient is assessed only once, at a random time between admission and discharge to the ICU/nursing ward, for a maximum of 1 day.
  The proportion of successful DeltaScan measurements, meaning the number of patients with a positive or negative test result in relation to the total number of patients tested with DeltaScan.
Repeatability of DeltaScan's Delirium Probability Score during three consecutive DeltaScan measurements | From date of study start until the date of study completion. Each patient is assessed only once, at a random time between admission and discharge to the ICU/nursing ward, for a maximum of 1 day.
  The variability of DeltaScan's Delirium Probability Score (on a scale from 1 (low probability of delirium) to 5 (high probability of delirium)) in patients scored as delirious, non-delirious and indeterminate across three measurements performed within a short time frame of 30 minutes. This will be done in a subsample of 30 delirious patients and 30 non-delirious patients.

OTHER OUTCOMES:
Change in positive and negative predictive values of DeltaScan between age subgroups on the ICU | The change in positive and negative predictive values between age groups is assessed through study completion. Each patient is assessed only once, at a random time between admission and discharge to the ICU/nursing ward, for a maximum of 1 day.
  Change in positive and negative predictive values of DeltaScan between ICU patients older than 60 years and patients 18 to 60 years old, in order to assess generalizability to younger patients.

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Numan T, van den Boogaard M, Kamper AM, Rood PJT, Peelen LM, Slooter AJC; Dutch Delirium Detection Study Group. Delirium detection using relative delta power based on 1-minute single-channel EEG: a multicentre study. Br J Anaesth. 2019 Jan;122(1):60-68. doi: 10.1016/j.bja.2018.08.021. Epub 2018 Oct 2. PMID 30579407
- [Background] van der Kooi AW, Zaal IJ, Klijn FA, Koek HL, Meijer RC, Leijten FS, Slooter AJ. Delirium detection using EEG: what and how to measure. Chest. 2015 Jan;147(1):94-101. doi: 10.1378/chest.13-3050. PMID 25166725